CLINICAL TRIAL: NCT00820742
Title: The Efficacy, Safety, and Tolerability of Pegaptanib Sodium in Filipino Patients With Neovascular Age-related Macular Degeneration: A Post Marketing Surveillance Study.
Brief Title: Efficacy, Safety, Tolerability of Pegaptanib Sodium (Macugen) in Filipino Patients With Neovascular Age Related Macular Degeneration.
Status: Withdrawn | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Other Study IDs: A5751025
Record Dates: First submitted 2009-01-08; First posted 2009-01-12 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: A5751025
MeSH Terms: interventions — pegaptanib

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Phase IV Post Marketing Surveillance Study: Open-label, observational study
  Interventions: Drug: Macugen

INTERVENTIONS:
Drug: Macugen — Intravitreous injection of Pegaptanib Sodium 3.47 mg/mL solution every 6 weeks

SUMMARY:
An open label, non-comparative, multicenter, non-interventional, post marketing surveillance study to evaluate the overall safety and tolerability of pegaptanib sodium(Macugen) in the treatment of Filipino patients with neovascular age-related macular degeneration based on incidence of adverse events and to evaluate the efficacy based on visual acuity, and the patient's and physician's overall satisfaction with tolerability and efficacy.

DETAILED DESCRIPTION:
Open-label, non-comparative, non-interventional study

ELIGIBILITY:
Inclusion Criteria:

* Must have at least one eye which was diagnosed with neovascular degeneration

Exclusion Criteria:

* Presence of other causes of choroidal neovascularization, including pathologic myopia (spherical equivalent of -8 diopters or more negative, or axial length of 25mm or more), ocular histoplasmosis syndrome, angioid streaks, choroidal rupture, multifocal choroiditis

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male of female 50 years and older, diagnosed with age-related macular degeneration
Enrollment: 0 (Actual)
Dates: Start 2008-02; Primary Completion 2009-05 (Estimated); Study Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events and serious adverse events | 12 months

SECONDARY OUTCOMES:
Mean change in visual acuity in the study eye at 6 months from baseline | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5751025&StudyName=Efficacy%2C%20safety%2C%20tolerability%20of%20Pegaptanib%20Sodium%20in%20Filipino%20patients%20with%20neovascular%20age%20related%20macular%20degeneration.